CLINICAL TRIAL: NCT07177079
Title: High-dose Ascorbate (HDA) in Combination With Azacitidine and Venetoclax (Aza/Ven) in Newly Diagnosed Acute Myeloid Leukemia (AML)
Brief Title: High-dose Ascorbate (HDA) in Combination With Standard of Care Azacitidine and Venetoclax in Acute Myeloid Leukemia (AML)
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Kittika Poonsombudlert (Other)
Responsible Party: Sponsor-Investigator, Kittika Poonsombudlert, Clinical Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202506290
Record Dates: First submitted 2025-09-09; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Azacitidine; venetoclax; Ascorbic Acid; Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- A. Standard of Care (azacitidine and venetoclax) (Active Comparator): Twelve patients will be randomized to Arm A.
  Interventions: Drug: Azacitidine; Drug: Venetoclax; Drug: Decitabine
- B. High-dose ascorbate administered concomitantly with azacitidine and venetoclax (Experimental): As this is the ﬁrst time high-dose ascorbate has been administered in combination with standard of care (azacitidine and venetoclax), the safety of the combination will be assessed in the ﬁrst 6 patients randomized to Arm B. These patients will continue with the expansion portion of the study, and an additional 6 patients will be added for a total of 12.
  Interventions: Drug: Azacitidine; Drug: Venetoclax; Drug: High-dose ascorbate; Drug: Decitabine

INTERVENTIONS:
Drug: Azacitidine — A chemotherapy drug known as a hypomethylating agent
Drug: Venetoclax — Targeted cancer therapy used to treat certain blood cancers. It specifically targets a protein called BCL-2 to trigger the self-destruction of cancer cells.
Drug: High-dose ascorbate — Administering vitamin C intravenously to achieve very high concentrations in the bloodstream. In contrast to low doses, which act as antioxidants, these pharmacological doses can function as a pro-oxidant, killing cancer cells while leaving healthy cells unharmed.
  Other Names: Vitamin C
  Arms: B. High-dose ascorbate administered concomitantly with azacitidine and venetoclax
Drug: Decitabine — Azacitidine may be substituted with decitabine 20 mg/m2 daily, on days 1-5, at PI discretion in the event of toxicity/drug supply shortage.

SUMMARY:
This is a randomized, open-label, Phase I clinical study with expansion. It will assess the safety and efficacy of high-dose ascorbate administered concomitantly with azacitidine and venetoclax in newly diagnosed AML.

DETAILED DESCRIPTION:
The purpose of this research study is to see if adding high dose ascorbate (vitamin c) intravenous infusion (IV) to the standard treatment regimen for AML (azacitidine/venetoclax or decitabine/venetoclax) is safe, and also to see if the addition of high dose ascorbate enhances the anti-AML impact of the azacitidine given with standard care.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥ 18 who are deemed unﬁt for intensive chemotherapy by meeting at least one of the following criteria:

  * age ≥ 75
  * Eastern Cooperative Oncology Group (ECOG) performance of 2-3
  * Severe cardiac disorder (e.g., congestive heart failure requiring treatment, ejection fraction ≤ 50%, or chronic stable angina)
  * Severe pulmonary disorder (e.g., DLCO ≤ 65% or FEV1 ≤ 65%)
  * Creatinine clearance < 45 mL/min
  * Hepatic disorder with total bilirubin > 1.5 times the upper limit of normal
  * Any other comorbidity that the investigators determine to be incompatible with intensive chemotherapy
* Newly diagnosed (non-APL) acute myeloid leukemia except those with cytogenetic/molecular abnormalities in the exclusion criteria
* Participants must have adequate organ function, deﬁned as:

  * Aspartate aminotransferase (AST/SGOT) and alanine aminotransferase (ALT/SGPT) ≤ 3.0 x upper limit of normal (ULN)
  * International normalized ratio (INR) < 1.5 x ULN and partial thromboplastin time (PTT) < 1.5 x ULN (patient could be eligible if they respond appropriately to correction with FFP or cryoprecipitate)
* Patients with a history of antecedent myelodysplasia (MDS) are eligible if they have not had prior chemotherapy/hypomethylating agent (e.g., azacitidine or decitabine). Prior exposure to other investigational agents could be considered at PI's discretion
* Patients who have developed therapy-related AML after prior radiation or chemotherapy for other malignancy(ies) are eligible if they have not been exposed to hypomethylating agent (e.g., azacitidine or decitabine) and/or venetoclax
* Patients presenting with marked leukocytosis (WBC > 25 k/mm3) should receive cytoreduction with hydroxyurea or cytarabine dose ≤ 1 g/m2 to mitigate the risk of tumor lysis syndrome before initiation of therapy with venetoclax
* For female participants of childbearing potential, a negative serum or urine pregnancy test (sensitivity of at least 25 mIU/mL) at screening
* Ability to understand and the willingness to sign a written informed consent document.
* Both male and female participants of childbearing potential agree to use an adequate method of contraception from screening through 6 months after the last dose of study treatment.

Exclusion Criteria

* Patients who have received prior therapy to treat their AML (except for cytoreductive hydroxyurea or cytarabine dose ≤ 1 g/m2 for hyperleukocytosis)
* Known hypersensitivity or allergy to ascorbate, azacitidine/decitabine, or venetoclax
* AML patients with the following cytogenetic/molecular aberrations are not eligible i. t(8;21)(q22;q22.1)/RUNX1::RUNX1T1 ii. inv(16)(p13.1q22) or t(16;16)(p13.1;q22)/ CBFB::MYH11 iii. bZIP in-frame mutated CEBPA without any adverse mutations iv. KMT2A rearrangement v. NPM1 or IDH1 or IDH2 or FLT3-ITD or FLT3-TKD mutation
* Patients with kidney disease needing dialysis, diabetic nephropathy, renal transplant recipients, and those with history of acute or chronic oxalate nephropathy
* Patients with primary hemochromatosis or transfusional iron overload as defined as persistently elevated Ferritin > 1000 ng/mL.
* Patients with type I or type II diabetes mellitus on treatment with short acting insulin who need at least a daily blood glucose monitoring test via finger stick
* Patients with a prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or eﬃcacy assessment of the investigational regimen
* Other major co-morbidities as determined unsuitable per the treating physician
* HIV-infection that is uncontrolled by anti-retroviral therapy. (HIV-infected patients on eﬀective anti- retroviral therapy with undetectable viral load within 6 months are eligible for this study)
* Patients with G6PD (glucose-6-phosphate dehydrogenase) deﬁciency
* Patients who are on warfarin or other strong CYP3A4 inducer/inhibitor and cannot have a drug substitution or who decline the drug substitution

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Phase I: Dose-limiting toxicities (DLTs) according to CTCAE version 5.0 | Days 1 through 28
  As this is the ﬁrst time high-dose ascorbate has been administered in combination with standard of care aza/ven, the safety of the combination will be assessed in the ﬁrst 6 patients randomized to Arm B. An initial DLT assessment will be made when 3 participants have been randomized to the Investigational Arm B and are evaluable for DLTs. If at most 1 out of 3 participants experience a DLT, an additional cohort of 3 participants will be evaluated for DLTs. If at most 1 out of 6 participants experience a DLT, the combination will be deemed safe. Should greater than or equal to 2 (≥2) out of 3 or 6 participants experience a DLT, the combination will be deemed unsafe, and accrual will be terminated.
Expansion: Composite complete remission rate defined as the proportion of patients with a complete remission (CR or CRi) | Three years from initiation of study
  The primary objective of the expansion is to estimate the composite complete remission rate defined as the proportion of patients with a complete remission (CR or CRi) by the end of study treatment for each arm separately.

CONTACTS AND LOCATIONS:
Overall Officials: Kittika Poonsombudlert, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Health Care, Iowa City, Iowa, United States